CLINICAL TRIAL: NCT06075719
Title: Stroke Research Initiative to Advance Equity
Acronym: STRIVE
Status: Not yet recruiting | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, M. Carter Denny, Principle Investigator, Medstar Health Research Institute
Other Study IDs: STUDY00006503
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stroke Survivor: Survivor of acute ischemic stroke or intracerebral hemorrhage in the last 6 weeks
- Caregiver: Primary caregiver of stroke survivor

SUMMARY:
1. Assess patient-centered outcomes (PCOs) amongst stroke survivors and their caregivers in the MedStar Health system longitudinally.

   i. Utilize a community advisory board (CAB) of stroke survivors and their caregivers to identify the patient-centered outcome(s) that they determine to be most important and valuable to assess based on their lived experiences.

   ii. Collect the chosen PCOs at multiple time points using an electronic survey tool (e.g. Qualtrics, Tonic or RedCap)
2. Evaluate the impact of social determinants of health (SDoH) and experiences of discrimination on the chosen PCOs.
3. Examine whether there are differences in long-term PCOs amongst stroke survivors from different racial and ethnic groups.

2.2 Hypothesis: We hypothesize that stroke survivors that come from historically marginalized populations, specifically African American and Latinos, will have lower patient-centered outcome scores overall as compared to their Caucasian counterparts. In addition, we hypothesize that the difference PCO scores between Caucasian and African American and Latino populations will be due in part to experienced discrimination and not SDoH alone.

.

ELIGIBILITY:
Stroke Survivor:

Inclusion Criteria:

≥ 18 years old Acute Ischemic Stroke (AIS) or Intracerebral Hemorrhage (ICH) patients that have been cared for in the MedStar Healthcare system AIS of ICH in the last six weeks Ability to communicate in English, Spanish, Amharic, Mandarin Chinese or French (most common languages in the greater Washington, DC area)

Exclusion Criteria:

Transient Ischemic Attack (TIA) or Subarachnoid Hemorrhage (SAH) Unable to complete required forms Life expectancy less than 6 months

Caregiver Inclusion Criteria Age ≥ 18 Self-identify as primary caregiver for the stroke survivor Ability to communicate in English, Spanish, Amharic, Mandarin Chinese, French

Exclusion Criteria Unable to complete study survey forms Life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke Survivors from the MedStar Health System and their Caregivers.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10 (Estimated); Primary Completion 2028-10 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Patient-Centered Outcome Measures | 5 years
  Assess patient-centered outcomes (PCOs) amongst stroke survivors and their caregivers in the MedStar Health System longitudinally.
  Stroke Impact Scale and the Modified Caregiver Strain Index

SECONDARY OUTCOMES:
Social Determinants of Health | 5 years
  Evaluate the impact of social determinants of health (SDoH) on the chosen PCOs.
Discrimination | 5 years
  Evaluate the impact of patient-reported experiences of discrimination on the chosen PCOs.